CLINICAL TRIAL: NCT06727110
Title: Dentin Caries and Polymer-induced Liquid Precursor System (PILP): Adult Safety Study
Brief Title: Polymer Induced Liquid Precursor (PILP) in Adults in With Dentin Caries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-40868
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- PILP Conditioner and Cement (Experimental): PILP conditioner and cement placement prior to tooth restoration.
  Interventions: Device: PILP Cement
- PILP Conditioner (Experimental): PILP conditioner application prior to tooth restoration.
  Interventions: Device: PILP Conditioner
- No intervention (No Intervention): Placement of traditional dental restoration without additional intervention.

INTERVENTIONS:
Device: PILP Cement — PILP cement liner.
  Arms: PILP Conditioner and Cement
Device: PILP Conditioner — PILP solution.
  Arms: PILP Conditioner

SUMMARY:
The goal of this clinical trial is to learn if polymer-induced liquid precursor (PILP) can be used safely to treat dentin caries (cavities) in adults. The main question it aims to answer is: Is PILP (conditioner or liner) safe in adult teeth with dental caries? Researchers will compare PILP to a placebo (a look-alike substance that contains no drug) to see if PILP safely treats cavities in teeth.

Participants will: 1) Have PILP or placebo applied to their tooth prior to the placement of a filling in the tooth, 2) Complete two telephone calls within three months of filling placement and 3) Visit the clinic at three months and six months after the placement of the filling.

DETAILED DESCRIPTION:
The proposed study is a first-in-human safety evaluation of Polymer-Induced Liquid Precursor (PILP)-releasing dental materials for the treatment of deep carious lesions in adult posterior teeth.

The study will enroll adult patients diagnosed with carious lesions involving the dentin. Participants will be randomly assigned to one of three intervention groups. The primary objective is to assess the safety of PILP application, with a hypothesis that PILP can be safely used without causing adverse events to the tooth or patient.

Participants will undergo a series of visits starting with a comprehensive screening and consent process, followed by the assigned dental procedure involving caries removal and restoration. Follow-up evaluations will occur at 48 hours, 1 month, 3 months, and 6 months post-procedure to monitor for any symptoms or adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged 18 to sixty-four
3. In good general health as evidenced by medical history (ASA 1 or 2)
4. With at least one posterior tooth with caries to dentin

   1. The tooth must have a pulpal diagnosis of pulpal health (no irreversible pulpitis or periapical radiolucency)
   2. The tooth should have no existing restorations
   3. The caries should be a Class I or class V single surface lesion
   4. The tooth should be planned for restoration with intra-coronal restoration (composite or RMGI restoration)
   5. The tooth should be deemed as needing a restoration based on ICDAS (International Caries Detection and Assessment System)

Exclusion Criteria: Known allergic reactions to components of the study device

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulpal response | Tooth vitality testing will occur approximatley 3 months and 6 months after placement of the restoration.
  Tooth vitality (pulpal response) after intervention.

SECONDARY OUTCOMES:
Dental pain/sensitivity | Tooth pain will be assessed at 48 hours, 1 month, 3 month and 6 months after placement of the restoration.
  The dental pain/sensitivity assessment will include Visual Analog Scale (VAS) for dental pain.
Gingival Inflammation | Gingival inflammation will be assed by intra-oral clinical exam at 3 and 6 months post restoration placement.
  Intra-Oral Assessment and Photographs will assess gingival inflammation (Löe-Silness gingival index).
Periapical status | A dental radiograph of the tooth will be take at 3 and 6 months post restoration placement.
  Dental radiographs will assess periapical status (periapical index)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Habelitz, PhD, Principal Investigator — Stefan Habelitz, PhD
Locations (1):
- University of California San Francisco, School of Dentistry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacino M, Girn V, Nurrohman H, Saeki K, Marshall SJ, Gower L, Saeed E, Stewart R, Le T, Marshall GW, Habelitz S. Integrating the PILP-mineralization process into a restorative dental treatment. Dent Mater. 2019 Jan;35(1):53-63. doi: 10.1016/j.dental.2018.11.030. Epub 2018 Dec 10. PMID 30545611